Project: Jejunal Ketogenesis and Type 2 Diabetes (But2)

Informed Consent Form

NCT05767177

February 09, 2023

## Jejunal Ketogenesis and Type 2 Diabetes

## CONSENT TO PARTICIPATE IN THE PROJECT

I HAVE RECEIVED ORAL AND/OR WRITTEN INFORMATION ABOUT THE STUDY AND HAVE HAD THE OPPORTUNITY TO ASK QUESTIONS. I GET TO KEEP THE WRITTEN INFORMATION.

- I AGREE TO PARTICIPATE IN THE PROJECT INTESTINAL KETOGENESIS POTENTIAL SIGNIFICANCE FOR TYPE 2 DIABETES?
- I AGREE TO MY SAMPLES BEING SAVED IN A BIOBANK IN THE MANNER DESCRIBED IN THE RESEARCH SUBJECT INFORMATION.

PLACE AND DATE SIGNATURE

NAME CLARIFICATION